CLINICAL TRIAL: NCT00107822
Title: An Open-Label Safety Study to Evaluate the Use of S-Caine™ Peel (Lidocaine 7% and Tetracaine 7% Cream) in Pediatric Patients Undergoing a Minor or Major Dermal Procedure
Brief Title: Safety Study of S-Caine Peel (Skin Numbing Cream) Before a Painful Dermatologic Procedure in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCP-47-05
Record Dates: First submitted 2005-04-08; First posted 2005-04-11 (Estimated); Last update posted 2005-10-06 (Estimated); Status verified 2005-10

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

INTERVENTIONS:
Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%)

SUMMARY:
The purpose of this study is to evaluate the safety of one treatment of S-Caine™ Peel (skin numbing cream) applied on healthy skin before a painful dermatologic procedure in children. This study will also evaluate how well the S-Caine™ Peel eases the pain of the procedure.

DETAILED DESCRIPTION:
The practice of dermatology is seeing a rise in the number of surgical and laser procedures as technological advances have expanded the number of conditions amenable to these evolving therapies. Skin biopsies, shave excisions, deep excisions, electro-surgical procedures, intralesional injections, and laser surgery are frequently performed by dermatologists on a daily basis. Some pain accompanies almost all of these procedures, and a local anesthetic is commonly used. Traditionally, intracutaneous injection of lidocaine (with or without epinephrine) has been the anesthetic of choice. However, patients undergoing these procedures are often afraid of needles and syringes and the pain associated with injections. As a result, topical anesthetic agents have been explored and developed as painless alternatives to injected anesthesia.

S-Caine™ Peel (lidocaine 7% and tetracaine 7% cream) consists of a new eutectic formulation of lidocaine and tetracaine. S-Caine Peel is a topical local anesthetic cream that forms a pliable peel on the skin when exposed to air. S-Caine Peel is not occluded during application.

The pain associated with medical procedures is often under-treated in children. Children often undergo painful procedures with little or no anesthetic, even when effective therapy is available. Reasons for not providing available therapy in children include concerns over adverse side effects, as well as the length of time necessary to provide adequate anesthesia. Recent guidelines strongly advocate for the proactive treatment of pain in children, including the pain associated with medical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 0 through 17 years of age.
* Patient requires a minor or major dermal procedure.
* Patient's legal guardian is able to read and understand a written informed consent and has signed and dated a written informed consent. The patient must provide assent whenever possible.

Exclusion Criteria:

* Patient has known allergies, contraindications or sensitivities to lidocaine, tetracaine, or other local anesthetics of the amide or ester type or to any components of the test materials.
* Patient has known active atopic dermatitis at the designated treatment site.
* Patient has damaged, denuded or broken skin at the designated treatment site.
* Patient is pregnant or breastfeeding.
* Patient has participated in an investigational study or clinical trial of an unapproved drug within the previous 30 days.
* Patient was born prematurely (less than 38 weeks).
* Patient has enrolled in any previous study involving S-Caine Peel.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80
Dates: Start 2005-04; Study Completion 2005-05

PRIMARY OUTCOMES:
To evaluate the safety of a single administration of S-Caine Peel in providing dermal anesthesia over intact skin before a minor and major dermal procedure in pediatric patients

SECONDARY OUTCOMES:
To evaluate the adequacy of anesthesia provided for minor and major dermal procedures

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - International Dermatology Research, Inc., Miami, Florida
  - Jacobi Medical Center, The Bronx, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee